CLINICAL TRIAL: NCT05213104
Title: Assessment of Flecainide to Lower the Patent Foramen Ovale Closure Risk of Atrial Arrhythmia or Tachycardia
Acronym: AFLOAT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fonds de Dotation ACTION (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP201110; 2021-002608-10 (EudraCT Number)
Record Dates: First submitted 2021-12-20; First posted 2022-01-28 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Patent Foramen Ovale; Atrial Arrhythmia; Cryptogenic Stroke
Keywords: cryptongenic stroke; Percutaneous Patent Foramen Ovale closure; randomized controlled trial; Patent Foramen Ovale; Atrial arrhythmia; Atrial Fibrillation; flecainide
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke; Atrial Fibrillation | interventions — Flecainide

STUDY DESIGN:
Intervention Model Description: randomized, controlled, open-label study with a blind evaluation of all the endpoints (PROBE design)
Who Masked: Outcomes Assessor
Masking Description: only outcomes assessor will be blinded to the study arm (PROBE design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 - Flecainide 150 mg 6 months (Experimental): Flecainide 150 mg 6 months in addition to standard of care
  Interventions: Drug: Flecainide
- group 2 - Flecainide 150 mg 3 months (Experimental): Flecainide 150 mg 3 months in addition to standard of care
  Interventions: Drug: Flecainide
- group 3 - no Flecainide (No Intervention): to receive no additional treatment (standard of care only).

INTERVENTIONS:
Drug: Flecainide — Flecainide 150 mg 6 months in addition to standard of care
  Other Names: Flecainide Acetate 150 MG
  Arms: group 1 - Flecainide 150 mg 6 months
Drug: Flecainide — Flecainide 150 mg 3 months in addition to standard of care
  Other Names: Flecainide Acetate 150 MG
  Arms: group 2 - Flecainide 150 mg 3 months

SUMMARY:
About 30% of ischemic strokes are cryptogenic. Patent Foramen Ovale (PFO) is present in about 25% of the general population. In cryptogenic strokes, PFO has been shown to be overrepresented and recent intervention studies have confirmed that PFO has a causal link with stroke. In patients with recent cryptogenic stroke, these randomized studies have shown at least 50%-reduction of recurrent neurological events after PFO percutaneous closure compared with medical therapy alone. At the The risk of AF reported in these studies in certainly largely underestimated as only symptomatic and recorded episodes of AF have been declared. Patients often report palpitations without a dia gnosis of AF made on the ECG or a Holter. Long term ECG monitoring provides more accurate data on AF incidence.

Administration of flecainide has been shown to be effective in preventing Atrial arrhythmia and may be useful in preventing these Atrial arrhythmia(AA) episodes after PFO closure.

To the knowledge of the investigators, there is no study assessing the efficacy of any antiarrhythmic drug in the prevention of AFafter PFO closure. AFLOAT will be the first randomized study to possibly validate flecainide to prevent Atrial arrhythmia in these patients.

DETAILED DESCRIPTION:
AFLOAT is a national, multicenter, randomized, controlled, open-label superiority study with a blind evaluation of all the endpoints (PROBE design).

The interventional phase is followed by an observational phase as long as the patient is implanted with the ICM during when only the data of the device will be collected.

Screening and selection occurs before the procedure of PFO closure and an inform consent form is signed.

During the procedure of PFO closure, a small ICM (CONFIRM RX, ABBOTT) providing a long-term monitoring is implanted to detect all AA episodes.

Immediately after PFO closure, patients are randomly assigned, in a 1:1:1 ratio, in 3 groups : flecainide (150 mg per day in a single sustained-release dose) for 6 months (in addition to standard of care), flecainide (150 mg per day in a single sustained-release dose) for 3 months (in addition to standard Clinical follow-up is conducted during hospitalization, at 3 months (M3) and 6 months (M6-end-of-interventionnal phase) after discharge. A contrast echocardiography is recommended between 1 and 6 months. Telemonitoring provides notifications in case of arrhythmic event.

An observational period in patients who will keep the ICM beyond the 6-month follow-up period. Atrial arrhythmia detection will be continued.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* They are candidates for a procedure of PFO closure, whatever the indication (secondary prevention of stroke, platypnoea, decompression illness…). The indication must have been confirmed by a multidisciplinary team as recommended by the Haute Autorité de Santé.
* They are affiliated to Social Security
* They have provided a signed written consent form ICM implantation and randomization will occur only in patients with successful PFO closure without any major complications

Exclusion Criteria:

* History of atrial arrhythmia (paroxysmal, persistent or permanent)
* Electrocardiographic of ventricular pre-excitation or bundle-branch block (QRS >120ms)
* Ischemic heart disease
* Dilated or hypertrophic cardiomyopathy
* A history of heart failure, severe valvular heart disease, left ventricular dysfunction (ejection fraction <50 percent)
* A long QT interval or Brugada syndrome
* The bradycardia-tachycardia syndrome (resting heart rate, ≤50 beats per minute, or repetitive sinoatrial blocks during waking hours)
* Documentation of previous episodes of second or third-degree atrioventricular block
* High heart rate at baseline > 100 bmp
* Renal insufficiency (Glomerular filtration rate estimated by the Cockroft and Gault formula <30ml/min/m2),
* Previous hypokalemia (potassium level <3 mmol per liter)
* Suspected or known pregnancy (woman of childbearing potential must undergo a pregnancy test)
* A known hypersensibility to flecainide or its excipients
* Contemporaneous enrollment in an interventional clinical trial
* Intended use of a prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with at least one episode of atrial arrythmia | within 3 months after PFO closure
  percentage of patients with at least one episode of symptomatic or asymptomatic atrial arrhythmia episodes (≥30s) recorded on long-term monitoring with an insertable cardiac monitor (ICM) during the 3 months after PFO closure Atrial arrhythmia is defined as any episode of AF, atrial flutter or atrial tachycardia that lasts 30 seconds or more, in accordance with the 2012 consensus statement from the Heart Rhythm Society and others

SECONDARY OUTCOMES:
percentage of patients with at least one episode of atrial arrythmia(AA) | between the 3-months and 6-months follow-up visits
  Percentage of patients with at least one episode of symptomatic or asymptomatic AA (≥30s) recorded on long-term monitoring with ICM between 3 and 6 months after PFO closure

OTHER OUTCOMES:
percentage of patients with AA≥6 min | within 3 months after PFO closure
  Percentage of patients with at least one episode of symptomatic or asymptomatic AA (≥6 min) recorded on long-term monitoring with ICM device during the 3 months after PFO closure
percentage of stroke or TIA | within 6 months after PFO closure
  Percentage of patients with at least one episode of fatal or non-fatal stroke or Transient Ischemic Attack (TIA) during the 3 and 6 months after PFO closure
Percentage of non-scheduled practitioner-consultation or hospitalization for any cardiovascular reason | within 6 months after PFO closure
  Percentage of patients with at least one episode of non-scheduled practitioner-consultation or hospitalization for any cardiovascular reason during the 3 and 6 months after PFO closure
All-cause mortality | within 6 months after PFO closure
  All-cause mortality during the 3 and 6 months after PFO closure
Rate of Flecainide-related adverse events | from the Day 0 (V0) to the 6 months follow-up visit (V2)
  Rate of Flecainide-related adverse events
Percentage of patients with at least one episode of symptomatic or asymptomatic AA | from Day 0 (V0) till the ICM explantation (up to 2.5 years)
  Percentage of patients with at least one episode of symptomatic or asymptomatic AA episodes (≥6 min) recorded on long-term monitoring with ICM device during the whole follow-up period until battery run out or ICM removal.

CONTACTS AND LOCATIONS:
Overall Officials: Giles MONTALESCOT, MD,PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Pitié Salpetrière, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauguel-Moreau M, Guedeney P, Dauphin C, Auffret V, Clerc JM, Marijon E, Elbaz M, Aldebert P, Beygui F, Abi Khalil W, Da Costa A, Macia JC, Elhadad S, Cayla G, Iriart X, Laredo M, Rolland T, Temmar Y, Gheorghiu ME, Brugier D, Silvain J, Hammoudi N, Duthoit G, Diallo A, Vicaut E, Montalescot G; ACTION Study Group. Flecainide to Prevent Atrial Arrhythmia After Patent Foramen Ovale Closure: AFLOAT Study, A Randomized Clinical Trial. Circulation. 2024 Nov 19;150(21):1659-1668. doi: 10.1161/CIRCULATIONAHA.124.071186. Epub 2024 Sep 2. PMID 39222035
- [Derived] Hauguel-Moreau M, Guedeney P, Dauphin C, Auffret V, Marijon E, Aldebert P, Clerc JM, Beygui F, Elbaz M, Khalil WA, Da Costa A, Macia JC, Elhadad S, Cayla G, Brugier D, Silvain J, Hammoudi N, Duthoit G, Vicaut E, Montalescot G; ACTION Study Group. Flecainide to prevent atrial arrhythmia after patent foramen ovale closure, Rationale and design of the randomized AFLOAT study. Eur Heart J Cardiovasc Pharmacother. 2024 May 4;10(3):184-189. doi: 10.1093/ehjcvp/pvad100. PMID 38216511